CLINICAL TRIAL: NCT06491940
Title: Comparison of the Role of Losartan Alone vs Hydrochlorothiazide Plus Losartan on Proteinuria in Diabetic Nephropathy Patients
Brief Title: Comparison of the Role of Losartan Alone vs Hydrochlorothiazide Plus Losartan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LosartanBVH
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Proteinuria
MeSH Terms: conditions — Proteinuria | interventions — Losartan; hydrochlorothiazide, losartan drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan group (Experimental): Patients will receive Losartan (LS) 50 mg per day.
  Interventions: Drug: Losartan
- Losartan + Hydrochlorothiazide (Experimental): Patients will be given losartan LS (50 mg per day) and Hydrochlorothiazide (HCTZ) 12.5 mg per day as a combination therapy.
  Interventions: Drug: Losartan + Hydrochlorothiazide

INTERVENTIONS:
Drug: Losartan — Patients will receives Losartan (LS) 50 mg per day.
  Arms: Losartan group
Drug: Losartan + Hydrochlorothiazide — Patients will be given Losartan LS (50 mg per day) and Hydrochlorothiazide (HCTZ) 12.5 mg per day as a combination therapy.
  Arms: Losartan + Hydrochlorothiazide

SUMMARY:
Losartan, an angiotensin II receptor blocker, has already been established as a treatment for diabetic nephropathy due to its ability to reduce blood pressure and mitigate the progression of kidney damage. However, the addition of a diuretic like hydrochlorothiazide may offer synergistic benefits in reducing proteinuria by addressing both the underlying renal pathology and potential volume overload in these patients. The current study aims at determining and comparing the role of losartan alone vs hydrochlorothiazide plus losartan in reducing proteinuria in diabetic nephropathy patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders with ≥18 years of age.
* Presence of proteinuria/albuminuria at time of screening.
* Creatinine clearance of 30 mL/min or higher.

Exclusion Criteria:

* A systolic blood pressure of 180 mm Hg or higher, a diastolic blood pressure of 110 mm Hg or higher.
* Presence of a second primary renal disease in addition to diabetic nephropathy.
* Patients with type 1 diabetes.
* A history of a cardiovascular or cerebrovascular event within 3 months before inclusion.
* Serum potassium of 6.0 mmol/L or higher.
* Transplantation or immunosuppressive treatment.
* Contraindication for the use of losartan or hydrochlorothiazide.
* Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of proteinuria | 4 months
  Efficacy will be labeled yes if reduction of proteinuria/albuminuria from the value before commencing treatment will be observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical department, Bahawal Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data will be shared with other researchers on a reasonable request.